CLINICAL TRIAL: NCT00318747
Title: Asthma Immunotherapy With a Ragweed Allergen Immunostimulatory Sequence Conjugate
Brief Title: Treatment of Ragweed-Allergic Asthma With an Immunostimulatory Drug
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ITN031AD
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Asthma; Allergy; Allergic Rhinitis; Rhinitis, Allergic, Seasonal
Keywords: Amb a 1-Immunostimulatory Oligodeoxyribonucleotide Conjugate; AIC; Amb a I Protein; Ragweed Allergy; Hay Fever; Wheeze; Immunotherapy; Tolerance; Immunostimulatory; Ragweed Season; Asthma; Asthmatics; Asthmatic
MeSH Terms: conditions — Asthma; Hypersensitivity; Rhinitis, Allergic; Rhinitis, Allergic, Seasonal; Respiratory Sounds

INTERVENTIONS:
Drug: Amb a 1-immunostimulatory oligodeoxyribonucleotide conjugate (AIC)

SUMMARY:
This study will test the effectiveness of an investigational treatment for patients with ragweed-induced asthma, sometimes called fall seasonal asthma. The treatment being tested is a series of anti-ragweed shots. The purpose of the study is to determine whether a short series of injections with Amb a 1-immunostimulatory oligodeoxyribonucleotide conjugate (AIC) can cause a long-lasting reduction in the symptoms of asthma that are caused by fall hay fever allergies.

DETAILED DESCRIPTION:
Ragweed allergy is a common trigger of asthmatic flare-ups in people with asthma. Individuals with ragweed allergy suffer increased asthma symptoms during the fall allergy season, which generally runs from August to November. These flare-ups can significantly impact an asthma patient's quality of life. AIC is an investigational medicine that combines special DNA sequences that can modify the way the immune system responds. In AIC, these sequences are linked to a piece of the ragweed pollen molecule (known as Amb a 1) that causes hay fever symptoms. Injections of AIC have been shown to change the way the immune system responds to ragweed pollen in both animals and humans in a way that may lead to reduced hay fever symptoms.

In a previous study, AIC was safe and well tolerated, and patients exhibited a decrease in allergy symptoms lasting up to 2 years after treatment on average. This study will evaluate whether short-term use of AIC during the spring can cause long-term immune tolerance to ragweed, reduce asthma symptoms, and decrease use of asthma medications for future allergy seasons.

During the 2007 fall ragweed allergy season, participants will be observed and be asked to keep a diary of their asthma symptoms and medication use. In the spring of 2008, participants will be randomly assigned to receive six weekly doses of either the experimental medicine or placebo. Participants will be observed again for the 2008 fall ragweed season. Another series of three weekly doses of the assigned study treatment will be given in spring 2009, with observation through the 2009 fall ragweed allergy season and possibly the 2010 season. During the observation periods, participants will be asked to track their asthma symptoms and medication use and report this information to study staff. Study visits will be weekly during the spring and biweekly during the ragweed season, with a maximum of 16 visits per year. Allergy and lung tests as well as blood and urine collection will occur at selected study visits; these tests are designed to measure the participants' immune response.

ELIGIBILITY:
Inclusion Criteria:

* History of asthma
* History of asthma medication use during the 2005 fall ragweed season
* Suspected ragweed allergy
* Positive laboratory tests for ragweed allergy

Exclusion Criteria:

* Received immunotherapy for ragweed or other allergens within the 5 years prior to study entry
* Received anti-IgE (omalizumab) within the year prior to study entry
* 3 or more courses of oral corticosteroids for asthma within the year prior to study entry
* Inpatient hospitalization for asthma within the 5 years prior to study entry
* History of respiratory failure or intubation for asthma
* Smoking within the 6 months prior to study entry
* Greater than 5 pack/year history of smoking
* Clinically significant acute or chronic illness
* Chronic immunodeficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2006-04; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change in average daily asthma medication use between the 2007 and 2008 ragweed seasons

SECONDARY OUTCOMES:
Effect of AIC on selected secondary clinical outcome measures
safety of AIC in this population
mechanisms through which AIC may induce tolerance to ragweed

CONTACTS AND LOCATIONS:
Overall Officials: David Broide, MD, Study Chair — University of California, San Diego; Peter Creticos, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Bernstein Clinical Research Center, University of Cincinnati, Cincinnati, Ohio
  - Optimed Research, Ohio State University, Columbus, Ohio
  - Pennsylvania State University, Hershey, Pennsylvania

REFERENCES:
- [Background] Simons FE, Shikishima Y, Van Nest G, Eiden JJ, HayGlass KT. Selective immune redirection in humans with ragweed allergy by injecting Amb a 1 linked to immunostimulatory DNA. J Allergy Clin Immunol. 2004 Jun;113(6):1144-51. doi: 10.1016/j.jaci.2004.03.003. PMID 15208597
- [Background] Tulic MK, Fiset PO, Christodoulopoulos P, Vaillancourt P, Desrosiers M, Lavigne F, Eiden J, Hamid Q. Amb a 1-immunostimulatory oligodeoxynucleotide conjugate immunotherapy decreases the nasal inflammatory response. J Allergy Clin Immunol. 2004 Feb;113(2):235-41. doi: 10.1016/j.jaci.2003.11.001. PMID 14767435
- See also: Click here for the Immune Tolerance Network Web site — http://www.immunetolerance.org
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/